CLINICAL TRIAL: NCT07134855
Title: Evaluating Care Pathways for Chronic Respiratory Diseases in Brazil
Brief Title: Mitigating Chronic Respiratory Disease Through the Lens of Multimorbidity (MARES3)
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Sponsor
Other Study IDs: UCL Worktribe 6981600; NIHR 303125 (Other Grant/Funding Number: UK NIHR (National Institute for Health and Care Research))
Record Dates: First submitted 2025-07-30; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma; Preserved Ratio Impaired Spirometry (PRISM)
Keywords: chronic obstructive pulmonary disease; asthma; multi-morbidity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to investigate how individuals attending primary healthcare (PHC) services in Brazil for treatment of non-communicable diseases (NCDs), identified there as having abnormal spirometry or as being at high risk for lung health problems (such as asthma and chronic obstructive pulmonary disease-COPD, collectively referred to as chronic respiratory disease (CRDs)) using the COLA-6 questionnaire, are able to access diagnostic testing and treatment.

The investigators will re-assess people diagnosed with abnormal spirometry in the MARES1 study (NCT07050823) or identified as being at high-risk for CRDs in the MARES2 study (NCT07093021). The estimated sample size is 309 from MARES1 and 164 from MARES2 for a total sample size of 473.

Qualitative interviews will be conducted with a diverse subsample of 30 participants to explore their experience accessing CRD diagnosis and treatment, including barriers and facilitators, while all participants will undergo basic data collection and spirometry.

DETAILED DESCRIPTION:
The investigators aim to investigate how individuals attending primary healthcare (PHC) services in Brazil for treatment of non-communicable diseases (NCDs), identified there as having abnormal spirometry or as being at high risk for lung health problems (such as asthma and chronic obstructive pulmonary disease-COPD, collectively referred to as chronic respiratory disease (CRDs)) using the COLA-6 questionnaire, are able to access diagnostic testing and treatment.

The study will be carried out in PHC services, including Basic Health Units (BHUs) and Family Health Units (FHUs), located in the municipalities of São Carlos and São Paulo, both in the state of São Paulo, Brazil.

Individuals are being followed up after participation in MARES1 study (NCT07050823) and MARES2 study (NCT07093021), and had been originally recruited from PHC services, including BHUs and FHUs, located in the municipalities of São Carlos and São Paulo, Brazil. People were recruited if they were attending a PHC service for care of a NCD.

At the research visit, all participants will be asked about access to care. In addition, all participants will have application of the CAAT questionnaire, and the ACQ-7 questionnaire for those with asthma, and all participants will have measurement of pre- and post-bronchodilator spirometry and Fraction of Exhaled Nitric Oxide (FeNO).

A semi-structured interviews will be conducted with a sample of 30 patients diagnosed with abnormal spirometry results: 10 with COPD, 10 with asthma, and 10 with PRISm or restriction. These face-to-face interviews will use open-ended questions, be audio-recorded, transcribed, and anonymized before analysis. Participants will be randomly selected to ensure diversity in gender, age, socioeconomic status, and employment background. The interview will explore how participants accessed healthcare services for diagnostic confirmation and treatment, and how this process affected their health status. Topics will include barriers and facilitators, how doubts were clarified, the type of education they received regarding the disease, diagnosis, and treatment, and whether any changes occurred in their lifestyle or routine following diagnosis or treatment.

The qualitative analysis of the interviews will follow Braun and Clarke, which consists of six phases: 1) Familiarization with the data set; 2) Coding; 3) Generation of initial themes; 4) Development and review of themes; 5) Refinement, definition and naming of themes; and 6) Writing. Descriptive statistics will be used to describe responses to questionnaires and lung function testing, including changes from the values recorded at recruitment to MARES1 and MARES2.

ELIGIBILITY:
Inclusion Criteria:

Participated in MARES1 and MARES2, which recruited people with non-communicable diseases attending primary healthcare services in Brazil, identified as being at high-risk for, or confirmed as having chronic respiratory diseases.

Exclusion Criteria:

* No consent to take part in MARES3.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a non-communicable disease and found to be at high risk for, or newly diagnosed with a chronic respiratory disease
Sampling Method: Non-Probability Sample
Enrollment: 473 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Barriers and facilitators to accessing care for those with newly diagnosed / suspected chronic respiratory disease in primary healthcare services in Brazil. | A single assessment visit conducted six months following diagnosis (participants from MARES1) / identification of being at high risk for chronic respiratory disease (participants from MARES2).
  Barriers and facilitators to accessing care for those with newly diagnosed / suspected chronic respiratory disease in primary healthcare services in Brazil, assessed at qualitative interviews.

SECONDARY OUTCOMES:
Spirometry | A single assessment visit conducted six months following diagnosis (participants from MARES1) / identification of being at high risk for chronic respiratory disease (participants from MARES2).
  Pre-and post bronchodilator spirometry
Disease Control Questionnaire | A single assessment visit conducted six months following diagnosis (participants from MARES1) / identification of being at high risk for chronic respiratory disease (participants from MARES2).
  Chronic Airways Assessment Test (CAAT) questionnaire
FeNO | A single assessment visit conducted six months following diagnosis (participants from MARES1) / identification of being at high risk for chronic respiratory disease (participants from MARES2).
  Fractional Exhaled Nitric Oxide
Disease Control Questionnaire | A single assessment visit conducted six months following diagnosis (participants from MARES1) / identification of being at high risk for chronic respiratory disease (participants from MARES2).
  ACQ-7 (Asthma Control Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: John R Hurst, PhD FRCP, Principal Investigator — University College London Hospitals; Renata G Mendes, DFisio, Principal Investigator — Federal University of Sao Carlos (UFScar), Brasil
Locations (2):
- Brazil (2):
  - Multiple primary care sites, São Carlos, São Paulo
  - Multiple primary care sites, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual responses from qualitative interviews.

REFERENCES:
- [Derived] Mendes RG, Leonardi NT, Castello-Simoes V, Kawakami DMO, Souza JVR, Schafauser-Segundo NS, Simoes RP, Pinto FG, Araujo GHG, da Silva MMC, Moriguchi CS, Franco FJBZ, Pires Di Lorenzo VA, Jordan R, Martins S, Siddharthan T, Al Sharmah S, Barber J, Hurst JR. Mitigating chronic respiratory disease through the lens of multimorbidity: the MARES mixed-methods study protocol. BMJ Open. 2026 Jan 16;16(1):e109950. doi: 10.1136/bmjopen-2025-109950. PMID 41545050